CLINICAL TRIAL: NCT02993328
Title: A Double-Blind, Randomized, Placebo Controlled Safety, Tolerability & Efficacy Trial Of A New Botanical Drug Product At One Dose Level For The Treatment Of Mild-To-Moderate Plaque Psoriasis In Adult Subjects
Brief Title: A Trial of a Botanical Drug Containing East Indian Sandalwood Oil (EISO) for Treatment of Plaque Psoriasis in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study location changed
Sponsor: Santalis Pharmaceuticals, Inc. (Industry)
Collaborators: Fremantle Dermatology (Other); ClinDatrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAN021-02
Record Dates: First submitted 2016-12-07; First posted 2016-12-15 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAN021 Serum (Experimental): SAN021 is a serum containing 10% East Indian Sandalwood Oil. It is packaged in an amber glass bottle with a dropper top. The dose is 5 drops per 1% BSA involvement twice daily.
  Interventions: Drug: SAN021 Serum
- SAN021 Placebo (Placebo Comparator): SAN021 Placebo is a serum that does not contain East Indian Sandalwood Oil however, does contain a synthetic sandalwood fragrance. It is packaged in an amber glass bottle with a dropper top. The dose is 5 drops per 1% BSA involvement twice daily.
  Interventions: Drug: SAN021 Placebo

INTERVENTIONS:
Drug: SAN021 Serum — SAN021 is a serum containing 10% East Indian Sandalwood Oil. It is packaged in an amber glass bottle with a dropper top. The dose is 5 drops per 1% BSA involvement twice daily.
  Other Names: Active
  Arms: SAN021 Serum
Drug: SAN021 Placebo — SAN021 Placebo is a serum that does not contain East Indian Sandalwood Oil however, does contain a synthetic sandalwood fragrance. It is packaged in an amber glass bottle with a dropper top. The dose is 5 drops per 1% BSA involvement twice daily.
  Other Names: Placebo Serum
  Arms: SAN021 Placebo

SUMMARY:
This trial will be a double-blind, single-center, randomized, placebo controlled study to evaluate the safety, tolerability, and efficacy of SAN021 study drug when administered for up to 42 days to adults between the ages of 18 to 65 years who have a clinical diagnosis of mild-to-moderate plaque psoriasis.

DETAILED DESCRIPTION:
Patients will enter the Screening Period once the informed consent and photographic consent process has been completed. Patients with mild-to-moderate plaque psoriasis, as defined by a Psoriasis Area and Severity Index (PASI) score between 2 and 12,36 appropriate for topical treatment that covers a minimum of 0.5% and a maximum of 10% BSA, in the permitted treatment areas, and who meet all of the inclusion and none of the exclusion criteria will be enrolled.

Once subject eligibility is confirmed and the screening procedures completed, all enrolled subjects will start the Treatment Period of the study. All enrolled subjects will receive either 10% SAN021 or placebo serum (randomized in a 2:1 ratio) with the first dose applied at the Day 1 Study Visit. Subjects will be instructed on how to apply the study medication twice daily for 42 days.

Subjects will return to the clinic for study-related assessments on Study Days 8, 15, 29 and a final visit on Day 43. On Study Day 50, subject will receive a Follow-up phone call and be queried for condition status since going off study.

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥18 but ≤65 years of age
2. Have a clinical diagnosis of mild-to-moderate plaque psoriasis, as defined by a Psoriasis Area and Severity Index (PASI) score between 2 and 12,36 appropriate for topical treatment that covers a minimum of 0.5% and a maximum of 10% Body Surface Area (BSA), in the permitted treatment areas.
3. Are willing to treat all psoriasis occurring in the permitted treatment areas with only SAN021
4. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events.
5. Are willing to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural or artificial) for the duration of the study.
6. Are willing to refrain from using any lotions, moisturizer, cleansers, cosmetics or creams, other than those issued as part of the study, on the treatment areas during the treatment period.
7. If female of childbearing potential, must be willing to practice an acceptable form of birth control for the duration of the study.
8. Are able to give written informed consent in a manner approved by the Institutional Review Board or Ethics Review Committee and comply with the requirements of the study.
9. Are willing to avoid participation in any other clinical trial for the duration of this study.
10. Are willing to refrain from treating restricted areas, which will be excluded from all assessments and Body Surface Area (BSA) calculation. These areas are as follows: head, neck, fingernails, toenails, soles of feet, and palms of hands, axillae, or intertriginous areas.

Exclusion Criteria:

1. Have spontaneously improving or rapidly deteriorating plaque psoriasis, or pustular psoriasis as determined by the Investigator.
2. Have been treated, with prescription medication for plaque psoriasis, with no improvement in condition, within 60 days prior to the Baseline visit.
3. Are pregnant, breast-feeding, or planning to become pregnant during the study.
4. Have any evidence of systemic cancer, squamous cell carcinoma, basal cell carcinoma, or any other confounding skin condition.
5. Are undergoing treatments with topical antipsoriatic drug products other than corticosteroids within 14 days prior to the Baseline Visit, and for therapy containing corticosteroids or retinoids within 28 days prior to Baseline Visit.
6. Have open sores or open lesions in the treatment area(s).
7. Have any condition that, in the opinion of the investigator, would confound the safety and/or efficacy assessments of plaque psoriasis.
8. Have participated in any interventional clinical trial in the previous 30 days.
9. Have a known sensitivity to any of the constituents of the test product including sensitivities to sandalwood oil, fragrances, or any member of the Compositae family of vascular plants (e.g., sunflowers, daisies, dahlias, etc.).
10. Have used, are using, or are planning to use immunosuppressive or immunomodulatory medication (i.e., biologics), including oral or parenteral corticosteroids.
11. Have a history of alcohol or illegal drug/substance abuse, or suspected alcohol or illegal drug/substance abuse in the past two years.
12. Plan to seek alternative treatment of any kind for their psoriasis, in the eligible treatment areas or otherwise, during the trial period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-10 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety measured by Adverse Events | Total from Baseline to Day 43
  Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug.
Number of patients reporting discomfort during or immediately following SAN021 application | Patient reported from Baseline to Day 43
  Tolerability will be based on the number of patients reporting discomfort during or immediately following application of SAN021.
Patients achieving a Physician's Global Assessment of "clear" or "almost clear" at any time-point from Baseline to day 43 of the study. | Any time-point from Baseline to Day 43
  The primary preliminary efficacy endpoint will be number of patients achieving a Physician's Global Assessment of "clear" or "almost clear" at any time-point during the 43 days of therapy.

SECONDARY OUTCOMES:
Patients achieving at least a one grade improvement in Physicians Global Assessment score at any time-point from Baseline to Day 43 of the study. | Any time-point from Baseline to Day 43
  Percentage of patients achieving at least a 1-grade improvement in Physicians Global Assessment score.
Patients achieving a Psoriasis Area and Severity Index Score Improvement ≥ 25% at any time-point from Baseline to Day 43 of the study. | Any time-point from Baseline to Day 43
  percentage of patients who have a ≥ 25% reduction in the Psoriasis Area and Severity Index (PASI) score at any time-point from Baseline to Day 43 of the study.
Patients achieving a two grade improvement in Physicians Global Assessment score at any time-point from Baseline to Day 43 of the study. | Any time-point from Baseline to Day 43 of the study
  percentage of patients achieving a 2-grade improvement in the Physicians Global Assessment score at any time-point from Baseline to Day 43 of the study.
Patients achieving a Psoriasis Area and Severity Index Score Improvement ≥50% at any time-point from Baseline to Day 43 of the study. | Any time-point from Baseline to Day 43 of the study.
  percentage of patients who have a ≥50% reduction in the Psoriasis Area Severity Index (PASI) score at any time-point from Baseline to Day 43 of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology West, Fremantle, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No